CLINICAL TRIAL: NCT00551577
Title: Prospective, Randomized Phase II Clinical Trial to Select Primary Chemotherapy With Carboplatin and Docetaxel in Patients With Advanced Ovarian Cancer Stage FIGO IIIC and IV
Brief Title: Neoadjuvant Chemotherapy With Carboplatin and Docetaxel in Patients With Advanced Ovarian Cancer-Prospective, Randomized Phase II Clinical Trial
Acronym: PRIMOVAR-1
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Bonn (Other)
Collaborators: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRIMOVAR-1
Record Dates: First submitted 2007-10-30; First posted 2007-10-31 (Estimated); Last update posted 2007-10-31 (Estimated); Status verified 2007-10

CONDITIONS: Ovarian Neoplasms
Keywords: Ovarian neoplasms,; Neoadjuvant Therapy,; Docetaxel,; Neoplasm, Residual
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasm, Residual | interventions — Neoadjuvant Therapy; Carboplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A1 (Active Comparator): 3 cycles of Carboplatin/Docetaxel (3-weekly) preoperative and 3 cycles of Carboplatin/Docetaxel (3-weekly) postoperative
  Interventions: Procedure: neoadjuvant chemotherapy (Carboplatin/Docetaxel)
- A2 (Experimental): 2 cycles of Carboplatin/Docetaxel (3-weekly) preoperative and 4 cycles of Carboplatin/Docetaxel (3-weekly) postoperative
  Interventions: Procedure: neoadjuvant chemotherapy (Carboplatin/Docetaxel)

INTERVENTIONS:
Procedure: neoadjuvant chemotherapy (Carboplatin/Docetaxel) — 3 cycles of Carboplatin/Docetaxel (3-weekly) preoperative and 3 cycles of Carboplatin/Docetaxel (3-weekly) postoperative
  Arms: A1
Procedure: neoadjuvant chemotherapy (Carboplatin/Docetaxel) — 2 cycles of Carboplatin/Docetaxel (3-weekly) preoperative and 4 cycles of Carboplatin/Docetaxel (3-weekly) postoperative
  Arms: A2

SUMMARY:
The purpose of this study is to evaluate response to neoadjuvant chemotherapy by imaging and observation of anatomical and biological indicators (i.e. ascites or continuous measurement of tumor marker CA 125). Furthermore the optimal number of preoperative administered cycles of combination chemotherapy with carboplatin and docetaxel should be determined.

ELIGIBILITY:
Inclusion Criteria:

* histological confirmed ovarian neoplasm
* Figo stage IIIC (2cm extrapelvic disease) or Figo IV
* more than 500 ml ascites volume (measured by sonography)
* age > 18 years old
* ECOG <= 2
* adequate hepatological, renal and haematological function
* informed consent

Exclusion Criteria:

* concomitant or previous malignant diseases
* debulking procedures on initial surgical approach
* existing peripheral sensoric neuropathy >= grade 2
* acute infections
* mental disorders, cerebral metastasis
* bowel obstruction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2003-03; Study Completion 2008-01 (Estimated)

PRIMARY OUTCOMES:
Preoperative reduction of ascites volume | preoperative: after 2nd or 3rd cycle of chemotherapy (3-weekly course)

SECONDARY OUTCOMES:
Evaluation of overall response, Evaluation of postoperative tumor size, Evaluation of perioperative morbidity and mortality, QOL | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Walther C Kuhn, Prof. MD, Principal Investigator — University of Bonn
Locations (2):
- Germany (2):
  - Department of Gynaecolgy and Obstetrics, University hopsital, Bonn, Bonn
  - Department of Gynaecology, University hospital, Hamburg, Hamburg

REFERENCES:
- [Derived] Polcher M, Rudlowski C, Friedrichs N, Mielich M, Holler T, Wolfgarten M, Kubler K, Buttner R, Kuhn W, Braun M. In vivo intratumor angiogenic treatment effects during taxane-based neoadjuvant chemotherapy of ovarian cancer. BMC Cancer. 2010 Apr 13;10:137. doi: 10.1186/1471-2407-10-137. PMID 20388201
- [Derived] Polcher M, Braun M, Friedrichs N, Rudlowski C, Bercht E, Fimmers R, Sauerwald A, Keyver-Paik MD, Kubler K, Buttner R, Kuhn WC, Hernando JJ. Foxp3(+) cell infiltration and granzyme B(+)/Foxp3(+) cell ratio are associated with outcome in neoadjuvant chemotherapy-treated ovarian carcinoma. Cancer Immunol Immunother. 2010 Jun;59(6):909-19. doi: 10.1007/s00262-010-0817-1. Epub 2010 Jan 20. PMID 20087581